CLINICAL TRIAL: NCT01575834
Title: A Multicenter, International, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Assess the Efficacy and Safety of Romosozumab Treatment in Postmenopausal Women With Osteoporosis
Brief Title: Efficacy and Safety of Romosozumab Treatment in Postmenopausal Women With Osteoporosis
Acronym: FRAME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20070337; 2011-001456-11 (EudraCT Number)
Record Dates: First submitted 2012-04-04; First posted 2012-04-12 (Estimated); Results first posted 2018-11-08 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Osteoporosis, Osteoporosis-Postmenopausal, Bone Diseases-Metabolic, Bone Diseases, Musculoskeletal Diseases
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis; Bone Diseases, Metabolic; Bone Diseases; Musculoskeletal Diseases | interventions — romosozumab; Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Romosozumab (Experimental): Participants received 210 mg romosozumab subcutaneous injections once a month for 12 months, followed by 60 mg denosumab subcutaneously once every 6 months for 24 months.
  Interventions: Drug: Romosozumab; Drug: Denosumab
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injections once a month for 12 months, followed by 60 mg denosumab subcutaneously once every 6 months for 24 months.
  Interventions: Drug: Placebo; Drug: Denosumab

INTERVENTIONS:
Drug: Romosozumab — Administered by subcutaneous injection once a month (QM)
  Other Names: AMG 785; EVENITY™
  Arms: Romosozumab
Drug: Placebo — Administered by subcutaneous injection once a month (QM)
  Arms: Placebo
Drug: Denosumab — Administered by subcutaneous injection once every 6 months (Q6M)
  Other Names: Prolia®

SUMMARY:
The purpose of this study is to determine if treatment with romosozumab is effective in preventing fractures in women with postmenopausal osteoporosis

ELIGIBILITY:
Inclusion Criteria:

- Postmenopausal women with osteoporosis, defined as low bone mineral density (BMD T-score at the total hip or femoral neck of ≤ -2.50)

Exclusion Criteria:

* BMD T-score of ≤ -3.50 at the total hip or femoral neck
* History of hip fracture
* Any severe or more than 2 moderate vertebral fractures, as assessed by the central imaging based on lateral spine x-rays
* Use of agents affecting bone metabolism
* History of metabolic or bone disease (except osteoporosis)
* Vitamin D insufficiency (vitamin D repletion and rescreening is permitted)
* Current hyper- or hypocalcemia
* Current, uncontrolled hyper- or hypothyroidism
* Current, uncontrolled hyper- or hypoparathyroidism

Ages: 55 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7180 (Actual)
Dates: Start 2012-03-15 (Actual); Primary Completion 2015-12-14 (Actual); Study Completion 2016-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (185):
- United States (25):
  - Research Site, Tucson, Arizona
  - Research Site, Laguna Hills, California
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, Santa Maria, California
  - Research Site, Walnut Creek, California
  - Research Site, Lakewood, Colorado
  - Research Site, Leesburg, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Plantation, Florida
  - Research Site, Tampa, Florida
  - Research Site, Gainesville, Georgia
  - Research Site, New Orleans, Louisiana
  - Research Site, Bethesda, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Albuquerque, New Mexico
  - Research Site, Asheville, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Mayfield, Ohio
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Denton, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Madison, Wisconsin
- Argentina (4):
  - Research Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Research Site, Mar del Plata, Buenos Aires
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Buenos Aires
- Australia (8):
  - Research Site, Maroubra, New South Wales
  - Research Site, St Leonards, New South Wales
  - Research Site, Herston, Queensland
  - Research Site, Keswick, South Australia
  - Research Site, Footscray, Victoria
  - Research Site, Geelong, Victoria
  - Research Site, Heidelberg West, Victoria
  - Research Site, Nedlands, Western Australia
- Belgium (7):
  - Research Site, Brussels
  - Research Site, Genk
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Lommel
  - Research Site, Yvoir
- Brazil (3):
  - Research Site, Curitiba, Paraná
  - Research Site, São Paulo, São Paulo
  - Research Site, São Paulo
- Canada (6):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Lachine, Quebec
  - Research Site, Québec, Quebec
- Colombia (4):
  - Research Site, Medellín, Antioquia
  - Research Site, Barranquilla, Atlántico
  - Research Site, Bogota, Cundinamarca
  - Research Site, Bogotá
- Czechia (11):
  - Research Site, Brno
  - Research Site, České Budějovice
  - Research Site, Havlíčkův Brod
  - Research Site, Klatovy
  - Research Site, Ostrava-Trebovice
  - Research Site, Pardubice
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Praha 11 - Chodov
  - Research Site, Uherské Hradiště
  - Research Site, Zlín
- Denmark (7):
  - Research Site, Aalborg
  - Research Site, Århus C
  - Research Site, Ballerup Municipality
  - Research Site, Glostrup Municipality
  - Research Site, Hvidovre
  - Research Site, Odense
  - Research Site, Vejle
- Dominican Republic (2):
  - Research Site, Santo Domingo, Nacional
  - Research Site, Santo Domingo
- Estonia (3):
  - Research Site, Pärnu
  - Research Site, Tallinn
  - Research Site, Tartu
- Germany (13):
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Dresden
  - Research Site, Frankfurt am Main
  - Research Site, Görlitz
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heinsberg
  - Research Site, Hellersdorf
  - Research Site, Leipzig
  - Research Site, Magdeburg
  - Research Site, Marburg
  - Research Site, Schkeuditz
- Hungary (7):
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Hévíz
  - Research Site, Szeged
  - Research Site, Zalaegerszeg
- India (6):
  - Research Site, Bangalore, Karnataka
  - Research Site, Mumbai, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Jaipur, Rajasthan
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Vellore, Tamil Nadu
- Japan (44):
  - Research Site, Anjyo-shi, Aichi-ken
  - Research Site, Urayasu-shi, Chiba
  - Research Site, Fukui-shi, Fukui
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Fukutsu-shi, Fukuoka
  - Research Site, Kitakyushu-shi, Fukuoka
  - Research Site, Kurume-shi, Fukuoka
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Chitose-shi, Hokkaido
  - Research Site, Ishikari-shi, Hokkaido
  - Research Site, Sunagawa-shi, Hokkaido
  - Research Site, Akashi-shi, Hyōgo
  - Research Site, Kako-gun, Hyōgo
  - Research Site, Toride-shi, Ibaraki
  - Research Site, Morioka, Iwate
  - Research Site, Takamatsu, Kagawa-ken
  - Research Site, Kirishima-shi, Kagoshima-ken
  - Research Site, Minamikyusyu-shi, Kagoshima-ken
  - Research Site, Atugi-shi, Kanagawa
  - Research Site, Sagamihara-shi, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Sendai, Miyagi
  - Research Site, Chiisagata-gun, Nagano
  - Research Site, Matsumoto-shi, Nagano
  - Research Site, Ueda-shi, Nagano
  - Research Site, Bungoono-shi, Oita Prefecture
  - Research Site, Osaka, Osaka
  - Research Site, Takatsuki-shi, Osaka
  - Research Site, Saga, Saga-ken
  - Research Site, Fujimi-shi, Saitama
  - Research Site, Matsue, Shimane
  - Research Site, Fujinomiya-shi, Shizuoka
  - Research Site, Kikugawa-shi, Shizuoka
  - Research Site, Tokushima, Tokushima
  - Research Site, Hachioji-shi, Tokyo
  - Research Site, Kiyose-shi, Tokyo
  - Research Site, Minato-ku, Tokyo
  - Research Site, Ōta-ku, Tokyo
  - Research Site, Setagaya-ku, Tokyo
  - Research Site, Shinagawa-ku, Tokyo
  - Research Site, Suginami-ku, Tokyo
  - Research Site, Toshima-ku, Tokyo
  - Research Site, Kofu, Yamanashi
- Latvia (2):
  - Research Site, Liepāja
  - Research Site, Riga
- Lithuania (3):
  - Research Site, Kaunas
  - Research Site, Klaipėda
  - Research Site, Vilnius
- Mexico (3):
  - Research Site, Mexico City, Mexico City
  - Research Site, Monterrey, Nuevo León
  - Research Site, Ciudad Obregón, Sonora
- New Zealand (2):
  - Research Site, Christchurch
  - Research Site, Grafton, Auckland
- Poland (7):
  - Research Site, Dabrowka Dopiewo
  - Research Site, Elblag
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Świdnik
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Romania (2):
  - Research Site, Bucharest
  - Research Site, Timișoara
- Spain (4):
  - Research Site, Barcelona, Catalonia
  - Research Site, Pozuelo de Alarcón, Madrid
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
- Switzerland (5):
  - Research Site, Bern
  - Research Site, Fribourg
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Zurich
- United Kingdom (7):
  - Research Site, Chorley
  - Research Site, Glasgow
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Northwood
  - Research Site, Reading

REFERENCES:
- [Background] Cosman F, Crittenden DB, Adachi JD, Binkley N, Czerwinski E, Ferrari S, Hofbauer LC, Lau E, Lewiecki EM, Miyauchi A, Zerbini CA, Milmont CE, Chen L, Maddox J, Meisner PD, Libanati C, Grauer A. Romosozumab Treatment in Postmenopausal Women with Osteoporosis. N Engl J Med. 2016 Oct 20;375(16):1532-1543. doi: 10.1056/NEJMoa1607948. Epub 2016 Sep 18. PMID 27641143
- [Background] Cosman F, Crittenden DB, Ferrari S, Khan A, Lane NE, Lippuner K, Matsumoto T, Milmont CE, Libanati C, Grauer A. FRAME Study: The Foundation Effect of Building Bone With 1 Year of Romosozumab Leads to Continued Lower Fracture Risk After Transition to Denosumab. J Bone Miner Res. 2018 Jul;33(7):1219-1226. doi: 10.1002/jbmr.3427. Epub 2018 May 17. PMID 29573473
- [Background] Chavassieux P, Chapurlat R, Portero-Muzy N, Roux JP, Garcia P, Brown JP, Libanati C, Boyce RW, Wang A, Grauer A. Bone-Forming and Antiresorptive Effects of Romosozumab in Postmenopausal Women With Osteoporosis: Bone Histomorphometry and Microcomputed Tomography Analysis After 2 and 12 Months of Treatment. J Bone Miner Res. 2019 Sep;34(9):1597-1608. doi: 10.1002/jbmr.3735. Epub 2019 Jun 24. PMID 31233639
- [Background] Cosman F, Crittenden DB, Ferrari S, Lewiecki EM, Jaller-Raad J, Zerbini C, Milmont CE, Meisner PD, Libanati C, Grauer A. Romosozumab FRAME Study: A Post Hoc Analysis of the Role of Regional Background Fracture Risk on Nonvertebral Fracture Outcome. J Bone Miner Res. 2018 Aug;33(8):1407-1416. doi: 10.1002/jbmr.3439. Epub 2018 May 11. PMID 29750828
- [Background] Lewiecki EM, Dinavahi RV, Lazaretti-Castro M, Ebeling PR, Adachi JD, Miyauchi A, Gielen E, Milmont CE, Libanati C, Grauer A. One Year of Romosozumab Followed by Two Years of Denosumab Maintains Fracture Risk Reductions: Results of the FRAME Extension Study. J Bone Miner Res. 2019 Mar;34(3):419-428. doi: 10.1002/jbmr.3622. Epub 2018 Dec 3. PMID 30508316
- [Background] Miyauchi A, Dinavahi RV, Crittenden DB, Yang W, Maddox JC, Hamaya E, Nakamura Y, Libanati C, Grauer A, Shimauchi J. Increased bone mineral density for 1 year of romosozumab, vs placebo, followed by 2 years of denosumab in the Japanese subgroup of the pivotal FRAME trial and extension. Arch Osteoporos. 2019 Jun 5;14(1):59. doi: 10.1007/s11657-019-0608-z. PMID 31168657
- [Background] Miyauchi A, Hamaya E, Yang W, Nishi K, Libanati C, Tolman C, Shimauchi J. Romosozumab followed by denosumab in Japanese women with high fracture risk in the FRAME trial. J Bone Miner Metab. 2021 Mar;39(2):278-288. doi: 10.1007/s00774-020-01147-5. Epub 2020 Oct 15. PMID 33057807
- [Background] McCloskey EV, Johansson H, Harvey NC, Lorentzon M, Shi Y, Kanis JA. Romosozumab efficacy on fracture outcomes is greater in patients at high baseline fracture risk: a post hoc analysis of the first year of the frame study. Osteoporos Int. 2021 Aug;32(8):1601-1608. doi: 10.1007/s00198-020-05815-0. Epub 2021 Feb 3. PMID 33537844
- [Background] Eriksen EF, Chapurlat R, Boyce RW, Shi Y, Brown JP, Horlait S, Betah D, Libanati C, Chavassieux P. Modeling-Based Bone Formation After 2 Months of Romosozumab Treatment: Results From the FRAME Clinical Trial. J Bone Miner Res. 2022 Jan;37(1):36-40. doi: 10.1002/jbmr.4457. Epub 2021 Nov 19. PMID 34633116
- [Background] Miller PD, Adachi JD, Albergaria BH, Cheung AM, Chines AA, Gielen E, Langdahl BL, Miyauchi A, Oates M, Reid IR, Santiago NR, Vanderkelen M, Wang Z, Yu Z. Efficacy and Safety of Romosozumab Among Postmenopausal Women With Osteoporosis and Mild-to-Moderate Chronic Kidney Disease. J Bone Miner Res. 2022 Aug;37(8):1437-1445. doi: 10.1002/jbmr.4563. Epub 2022 May 20. PMID 35466448
- [Background] Takada J, Dinavahi R, Miyauchi A, Hamaya E, Hirama T, Libanati C, Nakamura Y, Milmont CE, Grauer A. Relationship between P1NP, a biochemical marker of bone turnover, and bone mineral density in patients transitioned from alendronate to romosozumab or teriparatide: a post hoc analysis of the STRUCTURE trial. J Bone Miner Metab. 2020 May;38(3):310-315. doi: 10.1007/s00774-019-01057-1. Epub 2019 Nov 9. PMID 31707465
- [Background] Miyauchi A, Hamaya E, Nishi K, Tolman C, Shimauchi J. Efficacy and safety of romosozumab among Japanese postmenopausal women with osteoporosis and mild-to-moderate chronic kidney disease. J Bone Miner Metab. 2022 Jul;40(4):677-687. doi: 10.1007/s00774-022-01332-8. Epub 2022 May 31. PMID 35639174
- [Background] Eriksen EF, Boyce RW, Shi Y, Brown JP, Betah D, Libanati C, Oates M, Chapurlat R, Chavassieux P. Reconstruction of remodeling units reveals positive effects after 2 and 12 months of romosozumab treatment. J Bone Miner Res. 2024 Jul 23;39(6):729-736. doi: 10.1093/jbmr/zjae055. PMID 38640512
- [Background] Lane NE, Betah D, Deignan C, Oates M, Wang Z, Timoshanko J, Khan AA, Binkley N. Effect of Romosozumab Treatment in Postmenopausal Women With Osteoporosis and Knee Osteoarthritis: Results From a Substudy of a Phase 3 Clinical Trial. ACR Open Rheumatol. 2024 Jan;6(1):43-51. doi: 10.1002/acr2.11619. Epub 2023 Nov 20. PMID 37985218
- [Background] McClung MR, Betah D, Deignan C, Shi Y, Timoshanko J, Cosman F. Romosozumab Efficacy in Postmenopausal Women With No Prior Fracture Who Fulfill Criteria for Very High Fracture Risk. Endocr Pract. 2023 Sep;29(9):716-722. doi: 10.1016/j.eprac.2023.06.011. Epub 2023 Jul 4. PMID 37406858
- [Background] Cosman F, Oates M, Betah D, Timoshanko J, Wang Z, Ferrari S, McClung MR. Romosozumab followed by denosumab versus denosumab only: a post hoc analysis of FRAME and FRAME extension. J Bone Miner Res. 2024 Sep 2;39(9):1268-1277. doi: 10.1093/jbmr/zjae116. PMID 39041711
- [Derived] Lane J, Langdahl B, Stone M, Kurth A, Oates M, Timoshanko J, Wang Z, Libanati C, Cosman F. Romosozumab in patients who experienced an on-study fracture: post hoc analyses of the FRAME and ARCH phase 3 trials. Osteoporos Int. 2024 Jul;35(7):1195-1204. doi: 10.1007/s00198-024-07049-w. Epub 2024 Apr 4. PMID 38573517
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 222 centers in Europe, Central/Latin America, Asia, North America, and Australia/New Zealand.
  The first participant enrolled on 15 March 2012 and the last participant enrolled on 06 December 2013.
Pre-assignment Details: Participants were randomized 1:1 to receive either romosozumab 210 mg or matched placebo for the 12-month, double-blind, placebo-controlled period. Randomization was stratified by age (< 75 years, ≥ 75 years) and prevalent vertebral fracture (yes, no), as determined by site staff at randomization based on local reading of the spine X-ray.
Groups:
- Placebo/Denosumab: Participants received placebo subcutaneous injections once a month for 12 months, followed by 60 mg denosumab subcutaneously once every 6 months for 24 months.
- Romosozumab/Denosumab: Participants received romosozumab 210 mg subcutaneous injections once a month for 12 months, followed by 60 mg denosumab subcutaneously once every 6 months for 24 months.
Period: Overall Study
Arm/Group | Placebo/Denosumab | Romosozumab/Denosumab
Started | 3591 | 3589
Received Double-blind Treatment | 3582 (Six participants received a dose of romosozumab in error during the double-blind period.) | 3575
Completed Double-blind Period | 3205 | 3185
Completed 24-month Study Period | 3032 | 2994
Completed | 2892 (Completed 36-month study period) | 2851 (Completed 36-month study period)
Not Completed | 699 | 738
Not completed — Withdrawal by Subject | 352 | 390
Not completed — Death | 81 | 74
Not completed — Other | 70 | 70
Not completed — Adverse Event | 63 | 61
Not completed — Lost to Follow-up | 55 | 68
Not completed — Noncompliance | 52 | 27
Not completed — Administrative decision | 15 | 33
Not completed — Ineligibility Determined | 5 | 8
Not completed — Protocol Deviation | 4 | 3
Not completed — Requirement for Alternative Therapy | 2 | 4

BASELINE CHARACTERISTICS:
Population: The full analysis set consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Denosumab | Romosozumab/Denosumab | Total
Number analyzed (Participants) | 3591 | 3589 | 7180
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (6.9) | 70.9 (7.0) | 70.9 (7.0)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 757 | 768 | 1525
  ≥ 65 years | 2834 | 2821 | 5655
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3591 | 3589 | 7180
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1416 | 1427 | 2843
  Not Hispanic or Latino | 2175 | 2162 | 4337
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2052 | 2063 | 4115
  Asian | 441 | 425 | 866
  Black or African American | 74 | 77 | 151
  American Indian/Alaska Native | 63 | 64 | 127
  Native Hawaiian/Other Pacific Islander | 1 | 0 | 1
  Multiple | 59 | 60 | 119
  Other | 901 | 900 | 1801
Prevalent Vertebral Fracture Strata per Randomization [Count of Participants; unit: Participants] — Strata per randomization for prevalent fracture were based on local reading of baseline spine radiographs.
  Participants
    Yes | 205 | 204 | 409
    No | 3386 | 3385 | 6771
Age Strata per Randomization [Count of Participants; unit: Participants]
  < 75 years | 2471 | 2470 | 4941
  ≥ 75 years | 1120 | 1119 | 2239

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With New Vertebral Fracture Through Month 12
Description: New vertebral fractures occurred when there was ≥ 1 grade increase from the previous grade of 0 in any vertebra from T4 to L4 using the Genant semiquantitative scoring method.
  The Genant semiquantitative scoring method was based on assessment of x-rays according to the following scale:
  * Grade 0 (Normal) = no fracture;
  * Grade 1 (Mild) = mild fracture, 20 to 25% reduction in vertebral height (anterior, middle, or posterior);
  * Grade 2 (Moderate) = moderate fracture, 25 to 40% reduction in anterior, middle, and/or posterior height;
  * Grade 3 (Severe) = severe fracture, greater than 40% reduction in anterior, middle, and/or posterior height.
Time Frame: 12 Months
Population: Primary efficacy analysis set includes all participants who had a baseline and ≥ 1 postbaseline evaluation of vertebral fracture during the 12 months, including participants with missing baseline Genant scores whose first postbaseline spinal radiograph showed no fracture on the same vertebrae. Last observation carried forward imputation was used.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants received placebo subcutaneous injections once a month for 12 months.
- Romosozumab: Participants received romosozumab 210 mg subcutaneous injections once a month for 12 months.
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 3322 | 3321
percentage of participants | 1.8 | 0.5
Statistical Analysis 1: Comparison: Placebo vs Romosozumab; Test type: Superiority; p < 0.001, Regression, Logistic — A fixed-sequence testing procedure was used for multiplicity adjustment of the coprimary and a subset of secondary efficacy endpoints to maintain the overall significance level at 0.05; Based on logistic regression model adjusted for age and prevalent vertebral fracture stratification variables; p-value based on score test; Odds Ratio (OR) = 0.27, 95% CI 2-sided [0.15 to 0.47] — Values < 1 for odds ratio favor romosozumab

2. Primary Outcome: Percentage of Participants With New Vertebral Fracture Through Month 24
Description: as for outcome 1
Time Frame: 24 months
Population: Primary efficacy analysis set includes all participants who had a baseline and ≥ 1 postbaseline evaluation of vertebral fracture during the 24 months, including participants with missing baseline Genant scores whose first postbaseline spinal radiograph showed no fracture on the same vertebrae. Last observation carried forward imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Denosumab | Romosozumab/Denosumab
Number analyzed (Participants) | 3327 | 3325
percentage of participants | 2.5 | 0.6
Statistical Analysis 1: Comparison: Placebo/Denosumab vs Romosozumab/Denosumab; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.24, 95% CI 2-sided [0.15 to 0.39] — Values < 1 for odds ratio favor romosozumab

3. Secondary Outcome: Percentage of Participants With a Clinical Fracture Through Month 12
Description: Clinical fractures included clinical vertebral and nonvertebral fractures (excluding skull, facial, mandible, cervical vertebrae, thoracic vertebrae, lumbar vertebrae, metacarpus, finger phalanges, and toe phalanges) that were associated with signs and/or symptoms indicative of a fracture. Clinical vertebral fractures were included regardless of trauma severity or pathologic fractures; nonvertebral fractures associated with high trauma severity or pathologic fractures were excluded.
Time Frame: 12 Months
Population: Full analysis set; Last observation carried forward imputation (LOCF) was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 3591 | 3589
percentage of participants | 2.5 | 1.6
Statistical Analysis 1: Comparison: Placebo vs Romosozumab; Test type: Superiority; p = 0.008, Cox proportional hazards — [p-value comment as in outcome 1, analysis 1]; Cox proportional hazards model adjusting for age and prevalent vertebral fracture stratification variables; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.46 to 0.89] — Hazard ratio < 1 favors romosozumab

4. Secondary Outcome: Percentage of Participants With a Nonvertebral Fracture Through Month 12
Description: A nonvertebral fracture was defined as a fracture present on a copy of radiographs or other diagnostic images such as computerized tomography (CT) or magnetic resonance imaging confirming the fracture within 14 days of reported fracture image date recorded by the study site, and/or documented in a copy of the radiology report, surgical report, or discharge summary, excluding skull, facial, mandible, cervical vertebrae, thoracic vertebrae, lumbar vertebrae, metacarpus, finger phalanges, and toe phalanges. In addition, fractures associated with high trauma severity or pathologic fractures were excluded.
Time Frame: 12 Months
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 3591 | 3589
percentage of participants | 2.1 | 1.6
Statistical Analysis 1: Comparison: Placebo vs Romosozumab; Test type: Superiority; p = 0.096, Cox proportional hazards — [p-value comment as in outcome 1, analysis 1]; Cox proportional hazards model adjusting for age and prevalent vertebral fracture stratification variables; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.53 to 1.05] — Hazard ratio < 1 favors romosozumab

5. Secondary Outcome: Percentage of Participants With a Nonvertebral Fracture Through Month 24
Description: A nonvertebral fracture was defined as a fracture present on a copy of radiographs or other diagnostic images such as computerized tomography (CT) or magnetic resonance imaging confirming the fracture within 14 days of reported fracture image date as recorded by the study site, and/or documented in a copy of the radiology report, surgical report, or discharge summary, excluding skull, facial, mandible, cervical vertebrae, thoracic vertebrae, lumbar vertebrae, metacarpus, finger phalanges, and toe phalanges. In addition, fractures associated with high trauma severity or pathologic fractures were excluded.
Time Frame: 24 Months
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Denosumab | Romosozumab/Denosumab
Number analyzed (Participants) | 3591 | 3589
percentage of participants | 3.6 | 2.7
Statistical Analysis 1: Comparison: Placebo/Denosumab vs Romosozumab/Denosumab; Test type: Superiority; p = 0.057, Cox proportional hazards — [p-value comment as in outcome 1, analysis 1]; Cox proportional hazards model adjusting for age and prevalent vertebral fracture stratification variables; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.57 to 0.97] — Hazard ratio < 1 favors romosozumab

6. Secondary Outcome: Percentage of Participants With a Clinical Fracture Through Month 24
Description: as for outcome 3
Time Frame: 24 Months
Population: Full analysis set; LOCF imputation was used
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Denosumab | Romosozumab/Denosumab
Number analyzed (Participants) | 3591 | 3589
percentage of participants | 4.1 | 2.8
Statistical Analysis 1: Comparison: Placebo/Denosumab vs Romosozumab/Denosumab; Test type: Superiority; p = 0.096, Cox proportional hazards — [p-value comment as in outcome 1, analysis 1]; Cox proportional hazards model adjusting for age and prevalent vertebral fracture stratification variables; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.52 to 0.87] — Hazard ratio < 1 favors romosozumab

7. Secondary Outcome: Percentage of Participants With a Major Nonvertebral Fracture Through Month 12
Description: A major nonvertebral fracture was a subset of nonvertebral fractures including pelvis, distal femur (ie, femur excluding hip), proximal tibia (ie, tibia excluding ankle), ribs, proximal humerus (ie, humerus excluding elbow), forearm, and hip.
Time Frame: 12 Months
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 3591 | 3589
percentage of participants | 1.5 | 1.0
Statistical Analysis 1: Comparison: Placebo vs Romosozumab; Test type: Superiority; p = 0.096, Cox proportional hazards — [p-value comment as in outcome 1, analysis 1]; Cox proportional hazards model adjusting for age and prevalent vertebral fracture stratification variables; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.44 to 1.02] — Hazard ratio < 1 favors romosozumab

8. Secondary Outcome: Percentage of Participants With a Major Nonvertebral Fracture Through Month 24
Description: as for outcome 7
Time Frame: 24 Months
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Denosumab | Romosozumab/Denosumab
Number analyzed (Participants) | 3591 | 3589
percentage of participants | 2.8 | 1.9
Statistical Analysis 1: Comparison: Placebo/Denosumab vs Romosozumab/Denosumab; Test type: Superiority; p = 0.096, Cox proportional hazards — [p-value comment as in outcome 1, analysis 1]; Cox proportional hazards model adjusting for age and prevalent vertebral fracture stratification variables; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.49 to 0.91] — Hazard ratio < 1 favors romosozumab

9. Secondary Outcome: Percentage of Participants With a New or Worsening Vertebral Fracture Through Month 12
Description: A new or worsening vertebral fracture was identified when there was a ≥ 1 grade increase from the previous grade in any vertebra from T4 to L4.
Time Frame: 12 Months
Population: Primary efficacy analysis set includes all participants who had a baseline and ≥ 1 postbaseline evaluation of vertebral fracture during the 24 months, including participants with missing baseline Genant scores whose first postbaseline spinal radiograph showed no fracture on the same vertebrae. LOCF imputation was used
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 3322 | 3321
percentage of participants | 1.8 | 0.5
Statistical Analysis 1: Comparison: Placebo vs Romosozumab; Test type: Superiority; p = 0.096, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.28, 95% CI 2-sided [0.17 to 0.49] — Values < 1 for odds ratio favor romosozumab

10. Secondary Outcome: Percentage of Participants With a New or Worsening Vertebral Fracture Through Month 24
Description: as for outcome 9
Time Frame: 24 Months
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Denosumab | Romosozumab/Denosumab
Number analyzed (Participants) | 3327 | 3325
percentage of participants | 2.5 | 0.7
Statistical Analysis 1: Comparison: Placebo/Denosumab vs Romosozumab/Denosumab; Test type: Superiority; p = 0.096, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.26, 95% CI 2-sided [0.16 to 0.41] — Values < 1 for odds ratio favor romosozumab

11. Secondary Outcome: Percentage of Participants With a Hip Fracture Through Month 12
Description: Hip fractures were defined as a subset of nonvertebral fractures including fractures of the femur neck, femur intertrochanter, and femur subtrochanter.
Time Frame: 12 Months
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 3591 | 3589
percentage of participants | 0.4 | 0.2
Statistical Analysis 1: Comparison: Placebo vs Romosozumab; Test type: Superiority; p = 0.18, Cox proportional hazards — [p-value comment as in outcome 1, analysis 1]; Cox proportional hazards model adjusting for age and prevalent vertebral fracture stratification variables; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.22 to 1.35] — Hazard ratio < 1 favors romosozumab

12. Secondary Outcome: Percentage of Participants With a Hip Fracture Through Month 24
Description: as for outcome 11
Time Frame: 24 Months
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Denosumab | Romosozumab/Denosumab
Number analyzed (Participants) | 3591 | 3589
percentage of participants | 0.6 | 0.3
Statistical Analysis 1: Comparison: Placebo/Denosumab vs Romosozumab/Denosumab; Test type: Superiority; p = 0.12, Cox proportional hazards — [p-value comment as in outcome 1, analysis 1]; Cox proportional hazards model adjusting for age and prevalent vertebral fracture stratification variables; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.24 to 1.04] — Hazard ratio < 1 favors romosozumab

13. Secondary Outcome: Percentage of Participants With a Major Osteoporotic Fracture Through Month 12
Description: Major osteoporotic fractures included clinical vertebral fractures and fractures of the hip, forearm and humerus. Fractures associated with high trauma severity or pathologic fractures were excluded.
Time Frame: 12 Months
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 3591 | 3589
percentage of participants | 1.8 | 1.1
Statistical Analysis 1: Comparison: Placebo vs Romosozumab; Test type: Superiority; p = 0.012, Cox proportional hazards; Cox proportional hazards model adjusting for age and prevalent vertebral fracture stratification variables; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.40 to 0.90] — Hazard ratio < 1 favors romosozumab

14. Secondary Outcome: Percentage of Participants With a Major Osteoporotic Fracture Through Month 24
Description: as for outcome 13
Time Frame: 24 Months
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Denosumab | Romosozumab/Denosumab
Number analyzed (Participants) | 3591 | 3589
percentage of participants | 3.1 | 1.9
Statistical Analysis 1: Comparison: Placebo/Denosumab vs Romosozumab/Denosumab; Test type: Superiority; p = 0.002, Cox proportional hazards; Cox proportional hazards model adjusting for age and prevalent vertebral fracture stratification variables; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.46 to 0.84] — Hazard ratio < 1 favors romosozumab

15. Secondary Outcome: Percentage of Participants With Multiple New or Worsening Vertebral Fractures Through Month 12
Description: A new or worsening vertebral fracture was identified when there was a ≥ 1 grade increase from the previous grade in any vertebra from T4 to L4. A participant had multiple new or worsening vertebral fractures when there were ≥ 2 vertebrae from T4 to L4 with ≥ 1 grade increase from the previous grade. The multiple new or worsening vertebral fractures need not have occurred at the same visit.
Time Frame: 12 Months
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 3322 | 3321
percentage of participants | 0.3 | 0.03
Statistical Analysis 1: Comparison: Placebo vs Romosozumab; Test type: Superiority; p = 0.011, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.11, 95% CI 2-sided [0.01 to 0.87] — Values < 1 for odds ratio favor romosozumab

16. Secondary Outcome: Percentage of Participants With Multiple New or Worsening Vertebral Fractures Through Month 24
Description: as for outcome 15
Time Frame: 24 Months
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Denosumab | Romosozumab/Denosumab
Number analyzed (Participants) | 3327 | 3325
percentage of participants | 0.5 | 0.03
Statistical Analysis 1: Comparison: Placebo/Denosumab vs Romosozumab/Denosumab; Test type: Superiority; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.06, 95% CI 2-sided [0.01 to 0.44] — Values < 1 for odds ratio favor romosozumab

17. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density at the Lumbar Spine at Month 12
Description: Bone mineral density (BMD) was measured by dual-energy x-ray absorptiometry (DXA). DXA scans were analyzed by a central imaging center.
Time Frame: Baseline and Month 12
Population: Primary efficacy analysis set for BMD includes all randomized participants who had a baseline and ≥ 1 post-baseline evaluation at or before the time point under consideration in the study period; LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 3148 | 3151
percent change | 0.4 (0.1) | 13.1 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Romosozumab; The treatment comparison of BMD at the lumbar spine was analyzed using an analysis of covariance (ANCOVA) model which included treatment, age and prevalent vertebral fracture stratification variables, and baseline value of the endpoint, machine type and machine type-by-baseline value interaction; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 12.7, 95% CI 2-sided [12.4 to 12.9], Standard Error of Mean 0.1

18. Secondary Outcome: Percent Change From Baseline In Bone Mineral Density at the Lumbar Spine at Month 24
Description: as for outcome 17
Time Frame: Baseline and Month 24
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo/Denosumab | Romosozumab/Denosumab
Number analyzed (Participants) | 2877 | 2861
percent change | 5.5 (0.1) | 16.6 (0.1)
Statistical Analysis 1: Comparison: Placebo/Denosumab vs Romosozumab/Denosumab; [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 11.1, 95% CI 2-sided [10.8 to 11.4], Standard Error of Mean 0.1

19. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Total Hip at Month 12
Description: as for outcome 17
Time Frame: Baseline and Month 12
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 3210 | 3197
percent change | 0.3 (0.1) | 6.0 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Romosozumab; The treatment comparison of BMD at the total hip was analyzed using an ANCOVA model which included treatment, age and prevalent vertebral fracture stratification variables, and baseline value of the endpoint, machine type and machine type-by-baseline value interaction; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 5.8, 95% CI 2-sided [5.6 to 6.0], Standard Error of Mean 0.1

20. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Total Hip at Month 24
Description: as for outcome 17
Time Frame: Baseline and Month 24
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo/Denosumab | Romosozumab/Denosumab
Number analyzed (Participants) | 2918 | 2903
percent change | 3.2 (0.1) | 8.5 (0.1)
Statistical Analysis 1: Comparison: Placebo/Denosumab vs Romosozumab/Denosumab; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 5.3, 95% CI 2-sided [5.1 to 5.5], Standard Error of Mean 0.1

21. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Femoral Neck at Month 12
Description: as for outcome 17
Time Frame: Baseline and Month 12
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 3210 | 3197
percent change | 0.3 (0.1) | 5.5 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Romosozumab; The treatment comparison of BMD at the femoral neck was analyzed using an ANCOVA model which included included treatment, age and prevalent vertebral fracture stratification variables, and baseline value of the endpoint, machine type and machine type-by-baseline value interaction; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 5.2, 95% CI 2-sided [4.9 to 5.4], Standard Error of Mean 0.1

22. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Femoral Neck at Month 24
Description: as for outcome 17
Time Frame: Baseline and Month 24
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo/Denosumab | Romosozumab/Denosumab
Number analyzed (Participants) | 2918 | 2903
percent change | 2.3 (0.1) | 7.3 (0.1)
Statistical Analysis 1: Comparison: Placebo/Denosumab vs Romosozumab/Denosumab; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 4.9, 95% CI 2-sided [4.7 to 5.2], Standard Error of Mean 0.1

ADVERSE EVENTS:
Time Frame: Double-blind treatment period: 12 months; Overall study: 36 months
Description: Six participants randomized to placebo received a dose of romosozumab in error during the double-blind period. Therefore, these 6 participants were included in the romosozumab group (ie, as treated) for safety analyses.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- 12-Month Double-blind Period: Placebo: Participants received placebo subcutaneous injections once a month for 12 months
- 12-Month Double-blind Period: Romosozumab: Participants received romosozumab 210 mg subcutaneous injections once a month for 12 months.
- 36-Month Study Period: Placebo/Denosumab: Participants received placebo subcutaneous injections once a month for 12 months, followed by 60 mg denosumab subcutaneously once every 6 months for 24 months.
- 36-Month Study Period: Romosozumab/Denosumab: Participants received romosozumab 210 mg subcutaneous injections once a month for 12 months, followed by 60 mg denosumab subcutaneously once every 6 months for 24 months.
Arm/Group | 12-Month Double-blind Period: Placebo | 12-Month Double-blind Period: Romosozumab | 36-Month Study Period: Placebo/Denosumab | 36-Month Study Period: Romosozumab/Denosumab
Serious Adverse Events (participants affected / at risk) | 314/3576 | 344/3581 | 733/3576 | 728/3581
Other Adverse Events (participants affected / at risk) | 2059/3576 | 2019/3581 | 2434/3576 | 2463/3581
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 12-Month Double-blind Period: Placebo (N=3576) | 12-Month Double-blind Period: Romosozumab (N=3581) | 36-Month Study Period: Placebo/Denosumab (N=3576) | 36-Month Study Period: Romosozumab/Denosumab (N=3581)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 9 | 4
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Hypocoagulable state (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 4
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Pernicious anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 3 | 0 | 5 | 2
Acute myocardial infarction (Cardiac disorders) | 4 | 6 | 10 | 16
Adams-Stokes syndrome (Cardiac disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 3 | 3 | 5 | 7
Angina unstable (Cardiac disorders) | 3 | 6 | 9 | 10
Aortic valve disease mixed (Cardiac disorders) | 0 | 0 | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 1 | 2 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 6 | 18 | 17
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 2
Cardiac arrest (Cardiac disorders) | 1 | 1 | 3 | 2
Cardiac failure (Cardiac disorders) | 1 | 5 | 7 | 10
Cardiac failure acute (Cardiac disorders) | 1 | 1 | 4 | 2
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 5 | 3
Cardiac failure congestive (Cardiac disorders) | 4 | 7 | 8 | 10
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2 | 5 | 4
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 2 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 1
Cor pulmonale (Cardiac disorders) | 0 | 0 | 0 | 2
Coronary artery disease (Cardiac disorders) | 3 | 4 | 7 | 7
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 2 | 2
Heart valve incompetence (Cardiac disorders) | 1 | 0 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Low cardiac output syndrome (Cardiac disorders) | 0 | 0 | 0 | 1
Mitral valve prolapse (Cardiac disorders) | 0 | 0 | 1 | 0
Mitral valve stenosis (Cardiac disorders) | 1 | 0 | 2 | 1
Myocardial infarction (Cardiac disorders) | 2 | 2 | 9 | 8
Myocardial ischaemia (Cardiac disorders) | 4 | 3 | 7 | 3
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Paroxysmal atrioventricular block (Cardiac disorders) | 0 | 0 | 1 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 2 | 1 | 2 | 4
Stress cardiomyopathy (Cardiac disorders) | 1 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 3 | 0 | 5 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 1 | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 2 | 5 | 2
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Vestibular ataxia (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Goitre (Endocrine disorders) | 1 | 2 | 3 | 5
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 2 | 1
Primary hyperaldosteronism (Endocrine disorders) | 1 | 1 | 1 | 1
Age-related macular degeneration (Eye disorders) | 0 | 0 | 1 | 0
Angle closure glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Blindness unilateral (Eye disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 5 | 4 | 14 | 13
Cystoid macular oedema (Eye disorders) | 0 | 1 | 0 | 1
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Lens disorder (Eye disorders) | 0 | 0 | 1 | 0
Posterior capsule rupture (Eye disorders) | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 2 | 0
Retinal disorder (Eye disorders) | 0 | 0 | 1 | 0
Uveitis (Eye disorders) | 0 | 0 | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 2 | 0 | 3
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 9 | 10
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 3 | 1
Acute abdomen (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anal prolapse (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Coeliac disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Colitis ischaemic (Gastrointestinal disorders) | 1 | 1 | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 4 | 2 | 5
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Femoral hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fistula of small intestine (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 6 | 2
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Hernial eventration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Ileus (Gastrointestinal disorders) | 1 | 1 | 2 | 2
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 2 | 3 | 3
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1 | 3
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Pancreatic cyst (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatic cyst rupture (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatic fistula (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 1 | 6
Pancreatitis chronic (Gastrointestinal disorders) | 2 | 1 | 2 | 1
Peritoneal adhesions (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Reflux gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 1 | 2 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 3 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 3
Asthenia (General disorders) | 1 | 0 | 2 | 0
Chest pain (General disorders) | 1 | 3 | 3 | 4
Complication associated with device (General disorders) | 0 | 1 | 0 | 1
Death (General disorders) | 5 | 5 | 9 | 13
General physical health deterioration (General disorders) | 1 | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0 | 1
Medical device discomfort (General disorders) | 0 | 1 | 0 | 1
Mucosal dryness (General disorders) | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 1 | 3 | 2
Non-cardiac chest pain (General disorders) | 0 | 4 | 3 | 10
Oedema peripheral (General disorders) | 1 | 0 | 3 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Sudden death (General disorders) | 1 | 0 | 4 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 2 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholangitis sclerosing (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 3 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 3 | 6 | 5
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 2 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 8 | 5 | 11 | 12
Cholelithiasis obstructive (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 1 | 1
Hepatic cyst (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 1
Abdominal sepsis (Infections and infestations) | 0 | 0 | 2 | 0
Abscess (Infections and infestations) | 0 | 1 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 2
Amoebiasis (Infections and infestations) | 0 | 1 | 0 | 1
Amoebic colitis (Infections and infestations) | 1 | 0 | 1 | 0
Amoebic dysentery (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 2 | 1 | 7 | 4
Appendicitis perforated (Infections and infestations) | 1 | 0 | 1 | 2
Arthritis bacterial (Infections and infestations) | 1 | 1 | 1 | 1
Bacterial tracheitis (Infections and infestations) | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 4 | 3 | 9
Bronchitis bacterial (Infections and infestations) | 1 | 1 | 1 | 1
Bronchitis viral (Infections and infestations) | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 5 | 11 | 11
Chikungunya virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Chlamydial infection (Infections and infestations) | 0 | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium colitis (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 3
Cystitis (Infections and infestations) | 1 | 0 | 2 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 2 | 0
Dermatitis infected (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 3 | 1 | 6 | 3
Empyema (Infections and infestations) | 0 | 1 | 0 | 2
Encephalitis (Infections and infestations) | 0 | 0 | 1 | 0
Enterobacter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 2 | 3 | 3
Escherichia sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 3 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1
Gangrene (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 3 | 6
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1 | 1
Hepatitis B (Infections and infestations) | 0 | 0 | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1 | 0 | 1
Hepatitis viral (Infections and infestations) | 0 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 1
Infected dermal cyst (Infections and infestations) | 1 | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1 | 1 | 2
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 0 | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 2 | 0 | 2 | 1
Intestinal gangrene (Infections and infestations) | 0 | 0 | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 2
Lyme disease (Infections and infestations) | 0 | 0 | 1 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 2
Medical device site joint infection (Infections and infestations) | 0 | 0 | 1 | 0
Meningitis pneumococcal (Infections and infestations) | 0 | 1 | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0
Osteomyelitis chronic (Infections and infestations) | 2 | 0 | 2 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 1 | 0
Perichondritis (Infections and infestations) | 0 | 0 | 1 | 0
Perineal abscess (Infections and infestations) | 1 | 0 | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 1 | 0
Pharyngitis bacterial (Infections and infestations) | 0 | 1 | 0 | 1
Phlebitis infective (Infections and infestations) | 0 | 0 | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 10 | 19 | 37 | 44
Pneumonia bacterial (Infections and infestations) | 2 | 2 | 4 | 2
Pneumonia cryptococcal (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 2
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1
Pyelocystitis (Infections and infestations) | 0 | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 3 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 1
Pyometra (Infections and infestations) | 0 | 0 | 1 | 0
Pyonephrosis (Infections and infestations) | 0 | 0 | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 2
Sepsis (Infections and infestations) | 1 | 4 | 3 | 7
Septic shock (Infections and infestations) | 0 | 1 | 0 | 4
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 2
Skin infection (Infections and infestations) | 1 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 2 | 0 | 2
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Tick-borne viral encephalitis (Infections and infestations) | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1
Ureteritis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 7 | 4 | 14 | 17
Urinary tract infection bacterial (Infections and infestations) | 3 | 3 | 4 | 4
Urosepsis (Infections and infestations) | 1 | 0 | 2 | 2
Vaginitis bacterial (Infections and infestations) | 0 | 1 | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 1 | 0
Wound abscess (Infections and infestations) | 0 | 0 | 0 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Cataract operation complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 3 | 1 | 4 | 2
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Eyelid injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 6 | 7
Femoral neck fracture (Injury, poisoning and procedural complications) | 8 | 3 | 14 | 11
Femur fracture (Injury, poisoning and procedural complications) | 7 | 4 | 19 | 9
Fibula fracture (Injury, poisoning and procedural complications) | 4 | 4 | 8 | 7
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 2 | 3 | 6
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 8 | 8
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Internal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 4 | 2
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Postoperative adhesion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Postoperative delirium (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 1
Radial head dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 5 | 3 | 17 | 14
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 3 | 2
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Stoma site ischaemia (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 4 | 4 | 7 | 7
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 4 | 2 | 12 | 8
Uterine dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound evisceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood lactic acid increased (Investigations) | 0 | 0 | 0 | 1
Blood pressure decreased (Investigations) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 1 | 0 | 1 | 1
Body mass index increased (Investigations) | 0 | 0 | 1 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 1
Gastric pH decreased (Investigations) | 0 | 0 | 1 | 0
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0
Influenza B virus test positive (Investigations) | 1 | 0 | 1 | 0
Liver function test increased (Investigations) | 1 | 0 | 1 | 0
Transaminases increased (Investigations) | 1 | 1 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1 | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 3 | 4
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3 | 5 | 4
Hyponatraemic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoosmolar state (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Mineral metabolism disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 5 | 5
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4 | 4
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 5 | 3
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 15 | 6 | 27 | 21
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 5 | 4
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 10 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Acral lentiginous melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 8 | 2
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 4 | 2
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2 | 1
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Angiocentric lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2 | 6 | 7
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1
Benign neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Benign pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 4 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 11 | 8
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 2
Cervix carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 3
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 2
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Granular cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1 | 4
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3 | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 7 | 10 | 13
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant neoplasm of conjunctiva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 3
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neoplasm of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Oesophageal squamous cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 3 | 3
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Paget's disease of nipple (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Pancoast's tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 3
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Paranasal sinus benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 1
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 1
Rectal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3 | 1
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tracheal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0 | 1 | 0
Arachnoid cyst (Nervous system disorders) | 0 | 0 | 1 | 0
Basal ganglia stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 0
Brain stem ischaemia (Nervous system disorders) | 1 | 0 | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 0 | 0 | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 4 | 0
Cerebellar ischaemia (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebral haematoma (Nervous system disorders) | 0 | 1 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 3
Cerebral infarction (Nervous system disorders) | 1 | 0 | 2 | 0
Cerebral ischaemia (Nervous system disorders) | 2 | 1 | 2 | 3
Cerebrovascular accident (Nervous system disorders) | 7 | 4 | 9 | 14
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 1 | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 1 | 0 | 1 | 1
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Cervicogenic headache (Nervous system disorders) | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Dementia (Nervous system disorders) | 0 | 0 | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 1 | 0
Diabetic coma (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 2
Embolic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 3 | 1 | 5
Facial paralysis (Nervous system disorders) | 0 | 1 | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 1 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 2 | 3 | 3
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 3 | 0 | 4 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 1 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 1 | 1
Hypotonia (Nervous system disorders) | 0 | 1 | 1 | 1
Internal carotid artery kinking (Nervous system disorders) | 1 | 0 | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 2 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 9 | 13
Lacunar infarction (Nervous system disorders) | 0 | 0 | 2 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 2 | 2
Lumbosacral radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 1
Meralgia paraesthetica (Nervous system disorders) | 0 | 1 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Motor dysfunction (Nervous system disorders) | 0 | 0 | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 0 | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 1
Nerve root compression (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 1 | 0 | 1 | 0
Nystagmus (Nervous system disorders) | 1 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 1
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 0 | 0 | 0 | 1
Paresis (Nervous system disorders) | 0 | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 1 | 2
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Post-traumatic headache (Nervous system disorders) | 0 | 0 | 1 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 1 | 1 | 2
Sciatica (Nervous system disorders) | 0 | 0 | 5 | 1
Seizure (Nervous system disorders) | 0 | 1 | 1 | 3
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Stupor (Nervous system disorders) | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 3 | 4 | 7 | 9
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 4 | 6 | 13
Tremor (Nervous system disorders) | 0 | 1 | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1
Vascular encephalopathy (Nervous system disorders) | 1 | 0 | 2 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 1 | 0
Device dislocation (Product Issues) | 0 | 0 | 1 | 2
Device malfunction (Product Issues) | 0 | 0 | 1 | 0
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 1 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 1 | 2
Depression (Psychiatric disorders) | 4 | 1 | 6 | 3
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 2
Major depression (Psychiatric disorders) | 1 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 1
Personality change due to a general medical condition (Psychiatric disorders) | 1 | 0 | 2 | 0
Pseudodementia (Psychiatric disorders) | 1 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Schizophreniform disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0
Transient psychosis (Psychiatric disorders) | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 1 | 5
Acute prerenal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 2 | 0 | 2 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0
Hydrocalyx (Renal and urinary disorders) | 0 | 1 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 2 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 2 | 0
Renal infarct (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ureteric perforation (Renal and urinary disorders) | 1 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 3 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary tract inflammation (Renal and urinary disorders) | 0 | 1 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 2 | 0 | 2 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 2 | 0 | 3
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1 | 1 | 2
Pelvic haematoma (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 2
Urogenital prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 3 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 5 | 2 | 7
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 2
Vaginal haematoma (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Vaginal polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 2 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3 | 8
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 15 | 6 | 28 | 22
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6 | 9
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Granuloma annulare (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Activities of daily living impaired (Social circumstances) | 0 | 1 | 0 | 1
Immobile (Social circumstances) | 1 | 0 | 1 | 0
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 | 0 | 1 | 0
Cataract operation (Surgical and medical procedures) | 0 | 0 | 0 | 2
Hysterectomy (Surgical and medical procedures) | 0 | 1 | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 1 | 0
Osteosynthesis (Surgical and medical procedures) | 0 | 0 | 0 | 1
Pulmonary resection (Surgical and medical procedures) | 0 | 0 | 1 | 0
Rehabilitation therapy (Surgical and medical procedures) | 0 | 1 | 0 | 1
Scar excision (Surgical and medical procedures) | 0 | 1 | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0 | 2 | 1
Aortic thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 1
Arterial stenosis (Vascular disorders) | 0 | 1 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 2
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 3
Deep vein thrombosis (Vascular disorders) | 2 | 2 | 3 | 5
Dry gangrene (Vascular disorders) | 0 | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 5 | 8 | 12 | 15
Hypertensive crisis (Vascular disorders) | 0 | 2 | 2 | 6
Hypertensive emergency (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 2
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 2 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 4 | 3
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 2 | 0 | 2
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 1 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 1
Varicose ulceration (Vascular disorders) | 1 | 0 | 2 | 1
Varicose vein (Vascular disorders) | 1 | 0 | 3 | 1
Vascular insufficiency (Vascular disorders) | 0 | 0 | 1 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 12-Month Double-blind Period: Placebo (N=3576) | 12-Month Double-blind Period: Romosozumab (N=3581) | 36-Month Study Period: Placebo/Denosumab (N=3576) | 36-Month Study Period: Romosozumab/Denosumab (N=3581)
Constipation (Gastrointestinal disorders) | 162 | 138 | 210 | 189
Diarrhoea (Gastrointestinal disorders) | 133 | 111 | 191 | 182
Influenza (Infections and infestations) | 180 | 169 | 240 | 237
Nasopharyngitis (Infections and infestations) | 439 | 460 | 622 | 651
Upper respiratory tract infection (Infections and infestations) | 172 | 161 | 255 | 236
Urinary tract infection (Infections and infestations) | 142 | 130 | 263 | 244
Viral upper respiratory tract infection (Infections and infestations) | 227 | 206 | 263 | 230
Contusion (Injury, poisoning and procedural complications) | 122 | 102 | 204 | 179
Fall (Injury, poisoning and procedural complications) | 319 | 255 | 539 | 484
Arthralgia (Musculoskeletal and connective tissue disorders) | 434 | 468 | 663 | 668
Back pain (Musculoskeletal and connective tissue disorders) | 380 | 373 | 573 | 518
Muscle spasms (Musculoskeletal and connective tissue disorders) | 140 | 163 | 201 | 211
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 172 | 168 | 260 | 263
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 210 | 184 | 329 | 321
Pain in extremity (Musculoskeletal and connective tissue disorders) | 299 | 278 | 407 | 417
Dizziness (Nervous system disorders) | 158 | 154 | 216 | 228
Headache (Nervous system disorders) | 206 | 235 | 270 | 293
Cough (Respiratory, thoracic and mediastinal disorders) | 117 | 130 | 179 | 189
Hypertension (Vascular disorders) | 260 | 219 | 411 | 384

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.